CLINICAL TRIAL: NCT06515327
Title: Effects of Corticosteroid Use on Restoration of Spontaneous Circulation in Cardiac Arrest Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara Etlik City Hospital (Other Government); Etimesgut Military Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Corticosteroid Cardiac Arrest
Record Dates: First submitted 2024-07-09; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cardiopulmonary Arrest; Corticosteroids Adverse Reaction
Keywords: Cardiac Arrest, Corticosteroids Use,
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steroid Group: Patients using corticosteroids for any reason before cardiac arrest
- Non-Steroid Group: Patients not using corticosteroids and having cardiac arrest

SUMMARY:
We aim to investigate the effects of pre-arrest corticosteroid use for any reason on the time of return of spontaneous circulation in patients experiencing witnessed cardiac arrest, either in-hospital or out-of-hospital. Additionally, we plan to study the effects of corticosteroid use on post-ROSC administration of vasoactive agents, required dosage of vasoactive agents and number of vasoactive agents needed in order to reach targeted blood pressure levels.

DETAILED DESCRIPTION:
Patients will be collected from Etlik City Hospital Emergency Medicine Department. Patients presenting with witnessed cardiac arrest, either in-hospital or out-of-hospital, will be enrolled in our study.

Inclusion Criteria:

Age 18 and above Witnessed cardiac arrest

Exclusion Criteria:

Traumatic cardiac arrest Forensic cases Cardiac arrest secondary to ST-elevation myocardial infarction Patients in whom spontaneous circulation could not be achieved despite cardiopulmonary resuscitation lasting more than 20 minutes Patients with inaccessible past medical records or unknown medication history Patients without identification Unwitnessed cardiac arrest Pregnant patients

Patients will be divided into two groups:

The first group will consist of 23 patients who used corticosteroid medications for any reason before experiencing cardiac arrest.

The second group will consist of 23 patients who did not use corticosteroid medications before cardiac arrest.

Following successful cardiopulmonary resuscitation and restoration of spontaneous circulation, the following parameters will be recorded for both groups: need for vasopressor support, number of vasopressor agents used, maximum dose of vasopressor agent(s) required to maintain mean arterial pressure (MAP) >65 mmHg, duration of stay in intensive care unit/emergency department, mortality rate, length of hospital stay, patients' medical histories, age, and gender.

These parameters will be compared between the corticosteroid-using and non-using groups, and statistical analysis will be conducted to evaluate differences between the two groups

ELIGIBILITY:
Inclusion Criteria:

Age 18 and above Witnessed cardiac arrest

Exclusion Criteria:

Traumatic cardiac arrest Forensic cases Cardiac arrest secondary to ST-elevation myocardial infarction Patients in whom spontaneous circulation could not be achieved despite cardiopulmonary resuscitation lasting more than 20 minutes Patients with inaccessible past medical records or unknown medication history Patients without identification Unwitnessed cardiac arrest Pregnant patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients over the age of 18 with witnessed cardiac arrest
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
return of spontaneous circulation | 20 minutes after cardiac arrest
  patients with return of spontaneous circulation within 20 minutes of cardiopulmonary resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Obling LER, Beske RP, Meyer MAS, Grand J, Wiberg S, Mohr T, Damm-Hejmdal A, Forman JL, Frikke-Schmidt R, Folke F, Moller JE, Kjaergaard J, Hassager C. Effect of prehospital high-dose glucocorticoid on hemodynamics in patients resuscitated from out-of-hospital cardiac arrest: a sub-study of the STEROHCA trial. Crit Care. 2024 Jan 22;28(1):28. doi: 10.1186/s13054-024-04808-3. PMID 38254130
- [Background] Bagate F, Coppens A, Masi P, de Prost N, Carteaux G, Razazi K, Mekontso Dessap A. Cardiac and vascular effects of low-dose steroids during the early phase of septic shock: An echocardiographic study. Front Cardiovasc Med. 2022 Sep 26;9:948231. doi: 10.3389/fcvm.2022.948231. eCollection 2022. PMID 36225952
- [Background] Ullian ME. The role of corticosteriods in the regulation of vascular tone. Cardiovasc Res. 1999 Jan;41(1):55-64. doi: 10.1016/s0008-6363(98)00230-2. No abstract available. PMID 10325953